CLINICAL TRIAL: NCT04428775
Title: A Phase IIa, Randomized, Open-label, Multi-Center, Multi-Dose Study to Evaluate the Effects of ALZT-OP1a in Subjects With Mild-Moderate Stage Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Safety and Biomarker Study of ALZT-OP1a in Subjects With Mild-Moderate ALS Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: AZTherapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AZT-006
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; Lou Gehrig's disease; mild ALS; moderate ALS; mild to moderate ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Cromolyn Sodium

STUDY DESIGN:
Intervention Model Description: Two doses of ALZT-OP1a (cromolyn) are being evaluated in this study. Each dose of ALZT-OP1a (cromolyn) will be co-administered with a stable dose of ALS standard-of-care treatment as prescribed by their physician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (Low Dose) (Experimental): Group I (n=40) will receive treatment regimen of ALZT-OP1a (cromolyn) 17.1 mg/twice a day (bid) (total of 34.2 mg/day)
  Interventions: Drug: ALZT-OP1a (cromolyn)
- Group II (High Dose) (Experimental): Group II (n=40) will receive treatment regimen of ALZT-OP1a (cromolyn) 34.2 mg/bid (total of 68.4 mg/day)
  Interventions: Drug: ALZT-OP1a (cromolyn)

INTERVENTIONS:
Drug: ALZT-OP1a (cromolyn) — 1. Mast cell stabilizer
  2. Neuroinflammatory microglial modulator
  3. anti-inflammatory
  Other Names: Cromolyn; Cromolyn sodium; Sodium cromoglycate

SUMMARY:
This is a Phase IIa, randomized, open-label, multi-center, multi-dose study for subjects with mild to moderate ALS. The protocol is designed to determine whether ALZT-OP1a treatment will positively impact neuro-inflammatory biomarkers and slow down or arrest functional decline in subjects with mild to moderate ALS.

DETAILED DESCRIPTION:
This Phase IIa study is designed as a randomized, open-label, multi-center, multi-dose study for subjects with mild to moderate ALS. The study will evaluate 1) safety, 2) tolerability, 3) changes in physical function measured using the ALSFRS-R, 4) two doses of ALZT-OP1a in order to determine an optimal and effective dose that could positively impact neuro-inflammatory biomarkers, and 5) to demonstrate preliminary evidence if this treatment could potentially slow down or arrest functional decline in subjects with mild to moderate ALS.

Up to 80 evaluable subjects will be randomly assigned to one of two treatment groups: Group I (n=40) will consist of low dose ALZT-OP1a, administered via dry powder inhalation; OR Group II (n=40), which will consist of high dose ALZT-OP1a, administered via dry powder inhaler.

Subjects will dose for 12 weeks and will be asked to return to the site for scheduled visits and biomarker collection at Week 4, Week 8, and Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-75 years, both inclusive;
* Must provide written informed consent before any study related procedures;
* Should be capable to complete all trial related procedures, assessments and visits in the judgement of Investigator;
* Familial or sporadic ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria;
* Disease duration from ALS diagnosis ≤24 months;
* ALSFRS-R total score ≥ 36 at screening visit;
* ALSFRS-R Breathing sub-score should be ≥9 at the time of screening;
* ALSFRS-R Bulbar sub-score should be ≥9 at the time of screening;
* Peak inspiratory flow rate (PIFR) ≥ 100 L/minute;
* Forced vital capacity (FVC) >70% of predicted value;
* Participant must be receiving treatment with stable dose of standard of care treatment for ≥30 days prior to signing informed consent.

Exclusion Criteria:

* Subjects with bulbar-onset ALS;
* Any use of non-invasive ventilation (e.g., continuous positive airway pressure, non-invasive bi-level positive airway pressure or non-invasive volume ventilation) for any portion of the day, or mechanical ventilation via tracheostomy, or on any form of oxygen supplementation;
* Any other significant neurological disorder which can interfere with study assessments, e.g., significant cognitive impairment and/or clinical dementia;
* Significant psychiatric illness like schizophrenia, bipolar disorder etc. Subjects with depression can be included, only if the depression has been stable and no episode of major depression has occurred in past one year;
* Severe cardiac disease (e.g.,corrected QT interval > 500ms), Torsade de Pointes, evidence of significant heart failure (New York Heart Association [NYHA] Class 3 or greater, myocardial infarction or unstable angina in the 6 months prior to screening);
* Any moderate-to-severe pulmonary disease or difficulty taking inhaled drugs;
* Inability to tolerate the administration of an oral inhaled powder via dry powder inhaler (DPI);
* Has taken any investigational study drug within 30 days or five half-lives of the drug, whichever is longer, prior to dosing;
* Currently taking cromolyn, or has taken cromolyn, within the past 12 months;
* Allergy to cromolyn or cromolyn products, such as Intal®, Nasalcrom®, Opticrom®, Gastrocrom®, etc.;
* Taking inhaled protein products on a chronic basis (such as insulin, parathyroid hormone [PTH], etc.);
* Subjects who weigh 88 lb (40 kg) or less, or, body mass index (BMI) of <17.5 or >35.0 at screening;
* Moderate-to-severe liver disease: aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin concentrations >3 times the upper limit of normal; patients with hepatic diseases such as hepatic cirrhosis, hepatic cancer and active hepatitis
* Moderate-to-severe renal disease: creatinine clearance <45 mL/min/1.73 m2 (by Cockcroft-Gault calculation);
* Any clinically significant disorder or laboratory abnormality that, in the investigator's opinion, could interfere with the subject's participation in the study, place the subject at increased risk, or confound interpretation of the study results;
* Pregnant or breast-feeding females or sexually active females with childbearing potential, if no adequate contraceptive measures are used.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Plasma Biomarkers | up to 12 weeks
  To measure the effect of ALZT-OP1a treatment on selected plasma biomarkers in ALS patients.
  Candidate biomarkers in ng/mL include: Beta-tryptase, Beta-Hexosaminidase
  Candidate biomarkers in pg/mL include: CXCL1, interferon-y, interleukin (IL)-1a, IL-1b, IL-2, IL-5, IL-6, IL-8, IL-10, IL-15, IL-17, macrophage inflammatory protein (MIP)-1a, MIP-1b, monocyte chemoattractant protein (MCP)-1, neurofilament light protein (NfL), tumor necrosis factor (TNF)-a, and vascular endothelial growth factor (VEGF)

SECONDARY OUTCOMES:
Changes from baseline in ALS disease progression | up to 12 weeks
  Measured by ALS Functional Rating Scale-Revised (ALSFRS-R) - Questionnaire
Time to Event Requiring Respiratory Support | up to 12 weeks
  Measured by the time to event requiring full-time or nearly full-time respiratory support from baseline by treatment arm.
Changes from baseline in pulmonary function (forced vital capacity) | up to 12 weeks
  Measured by changes in forced vital capacity (FVC) in percent predicted value from baseline by treatment arm.
Changes from baseline in pulmonary function (peak inspiratory flow rate) | up to 12 weeks
  Measured by changes in peak inspiratory flow rate (PIFR) in liters per minute from baseline by treatment arm.
Incidence of adverse event (tolerability) related to ALZT-OP1a | up to 12 weeks
  Evaluated by number and percentage of unexpected adverse events by treatment arm.
Number of participants with abnormal vital signs | up to 12 weeks
  Measured by changes in systolic / diastolic blood pressure, pulse rate, respiratory rate, and body temperature from baseline by treatment arm.
  The data will also be presented in shift tables as within normal limits, clinically significant, not clinically significant.
Number of participants with abnormal physical or neurological examinations | up to 12 weeks
  Review of all body systems and changes evaluated for clinical significance from baseline by treatment arm.
  The data will also be presented in shift tables as within normal limits, clinically significant, not clinically significant.
Number of participants with abnormal electrocardiograms (ECGs) | up to 12 weeks
  Measured by changes in heart rate, PR interval, QRS complex, and QT interval from baseline by treatment arm.
  The data will also be presented in shift tables as within normal limits, clinically significant, not clinically significant.
Number of participants with treatment emergent clinically significant laboratory assessments | up to 12 weeks
  The abnormal values will be presented by treatment arm from baseline.
  The data will also be presented in shift tables as within normal limits, clinically significant, not clinically significant.
Changes from baseline in suicidal ideation and behavior | up to 12 weeks
  Measured by changes in Columbia Suicide Severity Rating Scale (C-SSRS) from baseline; minimum score: 0 maximum score: 10; lower values represent a better outcome.
The number of study dropouts due to serious, unanticipated treatment emergent adverse events | up to 12 weeks
  The dropouts will be presented by treatment arm from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David R. Elmaleh, PhD, Study Director — AZTherapies, Inc.
Locations (6):
- United States (6):
  - UCSD Altman Clinical and Translational Research Institute, La Jolla, California
  - Mayo Clinic, Jacksonville, Florida
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Granucci EJ, Griciuc A, Mueller KA, Mills AN, Le H, Dios AM, McGinty D, Pereira J, Elmaleh D, Berry JD, Paganoni S, Cudkowicz ME, Tanzi RE, Sadri-Vakili G. Cromolyn sodium delays disease onset and is neuroprotective in the SOD1G93A Mouse Model of amyotrophic lateral sclerosis. Sci Rep. 2019 Nov 27;9(1):17728. doi: 10.1038/s41598-019-53982-w. PMID 31776380